CLINICAL TRIAL: NCT04316611
Title: Evaluation of the Effectiveness of Potassium Chloride in the Management of Out-of-hospital Cardiac Arrest by Refractory Ventricular Fibrillation
Brief Title: Potassium Chloride in Out-of-hospital Cardiac Arrest Due to Refractory Ventricular Fibrillation
Acronym: POTACREH
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: As the inclusion period in the study has ended and regulatory authorizations have expired on 26/12/2023, with no inclusions conducted.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP180577; 2019-002544-24 (EudraCT Number)
Record Dates: First submitted 2020-02-07; First posted 2020-03-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Out-of-hospital Cardiac Arrest (OHCA)
Keywords: Out-of-hospital cardiac arrest (OHCA); Potassium chloride; Refractory ventricular fibrillation; External electric shock; Defibrillation; Amiodarone; Lidocaine
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Ventricular Fibrillation | interventions — Potassium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Potassium chloride (Experimental): Potassium chloride
  Interventions: Drug: Potassium chloride

INTERVENTIONS:
Drug: Potassium chloride — Direct intravenous injection (IVD) 20 mmol potassium chloride

SUMMARY:
The purpose of this study is to evaluate, in patients presenting with out-of-hospital cardiac arrest (OHCA) by ventricular fibrillation, refractory to 3 external electric shocks, the efficacy of a direct intravenous injection of 20 mmol KCl on their survival at hospital arrival.

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest (OHCA) has a poor prognosis, with an overall survival rate of about 5% at discharge. Shockable rhythm cardiac arrests (ventricular fibrillation (VF) and pulseless ventricular tachycardia) have a better prognosis.

In case of shockable rhythm, treatment is based on defibrillation, thereafter failure of 3 external electric shocks, on direct intravenous administration of 300 mg amiodarone, followed in case of ineffectiveness by an additional direct intravenous administration of 150 mg amiodarone. Lidocaine, which has long been used in this indication, is currently only recommended when amiodarone is unavailable or inefficient. Nevertheless, these 2 drugs, while they may be effective in converting refractory ventricular fibrillation to normal rhythm, have marked cardiodepressant effects (bradycardia, and/or negative inotropic effect) that persist after direct intravenous administration. This explains, at least partially, why a recent study did not show a significant difference in hospital discharge survival between amiodarone, lidocaine and placebo in patients presenting with OHCA by refractory ventricular fibrillation.

During surgical procedures under extracorporeal circulation, a cardioplegia solution is administered to interrupt cardiac activity and facilitate the surgical procedure. From a patho-physiological level, the mode of action of these solutions is based on a high concentration of potassium, which reduces the membrane resting potential of the myocytes. By extension, direct intravenous administration of 20 mmol potassium chloride (KCl) has been shown to convert ventricular fibrillation, resulting in a return to an hemodynamically efficient organized heart rate within a few minutes. The kalemia were at the upper limit of normal (5.5 mmol/l) 10 min after this injection, and normal at 20 min. A recent clinical case of a patient under extracorporeal circulation resuscitation, presenting with a refractory ventricular fibrillation, demonstrated the efficacy of direct intravenous injection of 3 g potassium chloride, resulting in a return to a sinus rhythm within a few minutes.

The immediate advantage of potassium chloride, compared to amiodarone (and also lidocaine), is the absence of cardiodepressant effect (bradycardia and/or hypotension) persisting after a while from the injection time. The mode of action of direct intravenous injection of potassium chloride to reduce ventricular fibrillation is indeed linked to the peak of hyperkalemia, whereas since the kalaemia are afterwards rapidly normalized in a few minutes, there is no persistent deleterious effect following this injection of potassium chloride. In addition, in the case of cardiac arrest, since the patient is already under continuous external cardiac chest compressions, no supplementary deleterious consequences related to this transient hyperkalemia are expected.

Direct intravenous injection of potassium chloride into a patient in out-of-hospital cardiac arrest with refractory ventricular fibrillation with 3 external electric shocks, instead of amiodarone, should interrupt this ventricular fibrillation and then allow a rapid return to an organized heart rhythm, and thus restore effective spontaneous cardiac activity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age 18 or over).
* Patient suffering from an outpatient cardiac arrest of presumed cardiac origin and presenting refractory ventricular fibrillation despite 3 external electric shocks.
* Patient with a health insurance plan.

Exclusion Criteria:

* Proven pregnancy.
* Major incompetent (patient under guardianship or curatorship).
* Patient who does not yet have a functional venous pathway after the 3 external electric shocks have been performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Survival at hospital admission | At hospital admission up to 1 day
  Survival (return of spontaneous circulation) at hospital admission

SECONDARY OUTCOMES:
Number of pre-hospital return of spontaneous circulation (ROSC) | Pre-hospital setting, up to 1 day
  Return of spontaneous circulation in pre-hospital setting
Time to pre-hospital return of spontaneous circulation (ROSC) | Pre-hospital setting, up to 1 day
  Time, in minutes, from cardiac arrest to return of spontaneous circulation in pre-hospital setting
Total pre-hospital epinephrine dose | Pre-hospital setting, up to 1 day
  Total epinephrine dose in mg administered in the pre-hospital setting
Total number of pre-hospital external electric shocks | Pre-hospital setting, up to 1 day
  Total number of external electric shocks delivered in the pre-hospital setting
Total number of persistent or recurrent shockable rhythm disorders | Pre-hospital setting, up to 1 day
  Total number of persistent or recurrent rhythm disorders requiring an external electric shock in pre-hospital setting
  Total number of persistent or recurrent rhythm disorders requiring an external electric shock in pre-hospital setting
  Total number of persistent or recurrent rhythm disorders requiring an external electric shock in pre-hospital setting
Heart rate at hospital admission | At hospital admission, up to 1 day
  Measurement of heart rate when the patient arrives on the hospital ward
Blood pressure at hospital admission | At hospital admission, up to 1 day
  Measurement of systolic and diastolic blood pressure when the patient arrives on the hospital ward
Survival with good neurological outcome (Cerebral Performance Category (CPC) 1 or 2)at hospital discharge | At hospital discharge, up to maximum 3 months
  Survival with a good neurological prognosis (CPC scores 1 and 2) at hospital discharge
Survival with good neurological outcome (Cerebral Performance Category 1 or 2)at 3 months | At 3 months
  Survival with a good neurological prognosis (CPC scores 1 and 2) at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Romain Jouffroy, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP - SAMU de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jouffroy R, Ecollan P, Chollet-Xemard C, Prunet B, Elie C, Treluyer JM, Vivien B. Evaluation of the effectiveness of potassium chloride in the management of out-of hospital cardiac arrest by refractory ventricular fibrillation: Study protocol of the POTACREH study. PLoS One. 2023 Apr 12;18(4):e0284429. doi: 10.1371/journal.pone.0284429. eCollection 2023. PMID 37043520